CLINICAL TRIAL: NCT04481321
Title: ENDOCHAP Monocentric Cohort: Clinical and Molecular Study of Endometriosis and Adenomyosis
Brief Title: Clinical and Molecular Study of Endometriosis and Adenomyosis
Acronym: ENDOCHAP
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: NI18108
Record Dates: First submitted 2020-07-17; First posted 2020-07-22 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: Endometriosis; Adenomyosis
Keywords: Endometriosis; Adenomyosis; pain; infertility; disease progressiveness
MeSH Terms: conditions — Endometriosis; Adenomyosis; Pain; Infertility | interventions — Biological Products; Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Peripheral blood, Vaginal and urinary swab, Endometriosis lesions,endometrial biopsies, Myometer biopsies, Peritoneal fluid, Follicular fluid biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with benign gynaecologic disease: Patients consulting for endometriosis, pelvic pain, abnormal uterine bleeding and/or infertility, or for a pelvic mass,
  Interventions: Biological: Biological/Vaccine

INTERVENTIONS:
Biological: Biological/Vaccine
  Other Names: Peripheral blood,; Vaginal and urinary swab; Endometriosis lesions,endometrial biopsies; Myometer biopsies; Peritoneal fluid; Follicular fluid biopsies

SUMMARY:
The purpose of this study is to determine whether endometriosis and adenomyosis are progressive diseases, in terms of symptoms (pain, abnormal uterine bleeding and infertility), anatomical lesions size, and recurrences. We also aimed to address molecular questions on immune dialogues between ectopic lesions and the eutopic endometrium, auto-immunity in endometriosis and adenomyosis and the role of the microbiota in their respective pathophysiologies.

DETAILED DESCRIPTION:
Endometriosis and adenomyosis are benign gynecological conditions which affect more than 10% of women, that typically cause pain and / or infertility, thereby exerting a negative impact on the patients' quality of life.

Although the pathogenesis of endometriosis and adenomyosis are controversial, both diseases are defined by the presence of endometrial tissue outside the uterine cavity. Endometriosis is a heterogeneous disease, with three phenotypes: superficial peritoneal endometriosis (SUP), ovarian endometrioma (OMA), and deep infiltrating endometriosis (DIE) The most widely accepted pathophysiological hypothesis for endometriosis is that of the implantation of ectopic endometrial cells following peritoneal reflux. Endometriosis can be associated with adenomyosis, also heterogeneous, characterized by the infiltration of endometrial tissue into the myometrium, presenting different forms: diffuse, focal or cystic.

Due to diseases heterogeneity, the diagnosis of endometriosis and adenomyosis is difficult and affected patients are subject to a long delay for appropriate management.

We hypothesize that the disease may be progressive in terms of symptoms (pain, abnormal uterine bleeding and infertility), anatomical lesions and recurrences. Furthermore, highlighting specific clinical and molecular markers would shorten the diagnostic time.

ELIGIBILITY:
Inclusion Criteria:

* Women of age between - 18 and 42 years old.
* In-service care for one of the pelvic pain and/or infertility, or for a pelvic mass.
* Having a radiological diagnosis made by a referral practitioner and/or operated in the department

Exclusion Criteria:

* HIV-positive women, HBV and HCV
* During pregnancy
* Having a cancer diagnosis
* Refusing to sign a consent.

Ages: 18 Years to 42 Years | Sex: Female
Age Groups: Adult
Study Population: Women of age between - 18 and 42 years old.
  * In-service care for one of the pelvic pain and/or infertility, or for a pelvic mass.
  * Having a radiological diagnosis made by a referral practitioner and/or operated in the department.
Sampling Method: Non-Probability Sample
Enrollment: 5300 (Estimated)
Dates: Start 2006-05 (Actual); Primary Completion 2040-06 (Estimated); Study Completion 2040-12 (Estimated)

PRIMARY OUTCOMES:
Pain scores (analog visual scale), quantification of uterine bleeding (number of towels or tampon/day/month) and live birth rates | 10 years
  Composite outcome
Changes in lesions or recurrences to imaging performed during the gynaecological follow-up of the patient | 10 years

SECONDARY OUTCOMES:
Pain scores (analog visual scale), quantification of uterine bleeding (number of towels or tampon/day/month) and live birth rates | 1 year
Pain scores (analog visual scale), quantification of uterine bleeding (number of towels or tampon/day/month) and live birth rates | 3 years
Pain scores (analog visual scale), quantification of uterine bleeding (number of towels or tampon/day/month) and live birth rates | 5 years
Pain scores (analog visual scale), quantification of uterine bleeding (number of towels or tampon/day/month) and live birth rates | 7 years
Delays between the onset of symptoms and post-operative or radiological histological diagnosis with specialized imaging (transvaginal ultrasound, endorectal ultrasound, magnetic resonance imagingI | 10 years
meeting specific criteria for endometriosis and adenomyosis lesions | 10 years
Association between clinical parameters of interrogation and clinical examination and the presence of endometriosis. | 10 years
Association between clinical parameters of interrogation and clinical examination and the presence of adenomyosis. | 10 years
Association between clinical data and the occurrence of the disease | 10 years
Creating a score on clinical diagnosis | 10 years
- Evaluation of individualized management: comparison between different management strategies on pain scores (analog visual scale), pregnancy-conception desire delay, live birth rate | 10 years
Serum dosage of circulating antibodies before and after surgical treatment of lesions | 10 years
Metabolic pathway exploration in adenomyosis lesions | 10 years
Study of the presence of autoantibodies in cases of endometriosis and adenomyosis | 10 years
Establish a genotype/phenotype correlation of the disease (endometriosis and adenomyosis) | 10 years
To study the natural history of deep endometriosis lesions and analysis of focused invasion processes, epithelio-mesenchymatous transitions, and fibrogenesis using molecular biology techniques | 10 years
Characterization of the microbiota in urine and vaginal samples. | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Louis Marcellin, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Port Royal, hospital cochin, Paris, France

IPD SHARING:
Plan to Share IPD: No